CLINICAL TRIAL: NCT01758289
Title: A Prospective, Multicenter, Six-Month Study on the Effectiveness, Safety and Impact on Health Related Quality of Life (HRQoL) and Depression Symptoms of Paricalcitol Administered to Venezuelan Patients With Chronic Kidney Disease (Stage V) Who Are on Hemodialysis
Brief Title: Post Marketing Observational Study on Paricalcitol IV Administered to Venezuelan Patients
Status: Terminated | Type: Observational
Why Stopped: Changes in country regulation
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-785
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Kidney Disease Stage V; Hemodialysis
Keywords: Venezuelan Patients; Depressive Symptoms; Health Related Quality of Life
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Paricalcitol IV: Eligible participants with diagnosis of chronic kidney disease stage V undergoing hemodialysis, treated with paricalcitol IV per routine clinical practice according to prescribing information approved in Venezuela and clinical criteria.

SUMMARY:
This study was designed to evaluate the effectiveness, safety, and impact on quality of life when paricalcitol (Zemplar® intravenous [IV]) is administered in Venezuelan patients on hemodialysis who are at risk of developing secondary hyperparathyroidism associated with stage V chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years old with documented diagnosis of stage V chronic kidney disease, on hemodialysis at study baseline
* Subjects who have been previously treated with vitamin D or its metabolites or naïve to paricalcitol
* Subjects in whom the use of paricalcitol is clinically indicated and documented by applicable and routine standard of healthcare (i.e. laboratory assessments and clinical evaluations) according to the criteria of the attending physician and in accordance with the approved label of the product in Venezuela
* Subjects that provide written informed consent form stating his/her authorization and willingness to participate in the study and allowing the use and discussion of his/her personal and/or health information before entering the study
* Female subjects with reproductive potential must use an approved contraceptive method (intrauterine device, birth control pills or barrier device) during and for three (03) months after discontinuation of treatment

Exclusion Criteria:

* Subjects with severe hyperparathyroidism (parathyroid hormone [PTH] > 3000 pg/mL)
* Subjects with hypercalcemia, adjusted according to serum albumin, hyperphosphatemia, or subjects with calcium-phosphorus product (Ca x P) ≥ 70
* Known hypersensitivity and/or toxicity of vitamin D, its metabolites and/or other components of Zemplar® IV (paricalcitol)
* Subjects who have participated in clinical trials within 30 days before the start of the study or who are currently enrolled in a clinical trial or under treatment with any investigational product
* Subjects who cannot tolerate or cannot take phosphate binders that do not contain calcium and/or aluminum
* Subjects who in the opinion of the investigator, for any reason (including medical reasons) are not eligible and/or appropriate for therapy with synthetic analogs of vitamin D and/or unwilling to complete the study visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was conducted in 8 hemodialysis units distributed in Venezuela.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanine Obage, MD, Study Chair — Abbott
Locations (8):
- Venezuela (8):
  - Site Reference ID/Investigator# 96757, Acarigua
  - Site Reference ID/Investigator# 96766, Barquisimeto
  - Site Reference ID/Investigator# 96768, Caracas
  - Site Reference ID/Investigator# 96760, Maracaibo
  - Site Reference ID/Investigator# 96761, Maracaibo
  - Site Reference ID/Investigator# 96770, Miranda
  - Site Reference ID/Investigator# 96763, Monagas
  - Site Reference ID/Investigator# 96765, Naguanagua

RESULTS

PARTICIPANT FLOW:
Groups:
- Paricalcitol IV: Participants with a diagnosis of chronic kidney disease stage V undergoing hemodialysis were treated with paricalcitol intravenous (IV) per routine clinical practice, according to prescribing information approved in Venezuela and clinical criteria.
Period: Overall Study
Arm/Group | Paricalcitol IV
Started | 105
Completed | 52
Not Completed | 53
Not completed — Premature Study Termination | 44
Not completed — Adverse Event | 9

BASELINE CHARACTERISTICS:
Groups:
- Paricalcitol IV: Participants with a diagnosis of chronic kidney disease stage V undergoing hemodialysis were treated with paricalcitol IV per routine clinical practice, according to prescribing information approved in Venezuela and clinical criteria.
Arm/Group | Paricalcitol IV
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] — Missing data of one (1) participant, for whom age (years) was not reported.
  years | 53.00 (13.90)
Sex/Gender, Customized [Number; unit: participants]
  Female | 37
  Male | 67
  Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving at Least a 30% Reduction From Baseline in the Levels of Parathyroid Hormone (PTH) at the Final Study Visit
Time Frame: Baseline Week 1 (Study Visit 1) to Week 24 (Final Study Visit)
Population: Participants with valid PTH values at Baseline and Final Study Visit.
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol IV
Number analyzed (Participants) | 50
percentage of participants | 62

2. Secondary Outcome: Percentage of Participants With Hypercalcemia, Hyperphosphatemia and Elevations of Calcium-Phosphate Product (Ca x P) at Baseline, Week 12, and Week 24
Description: Hypercalcemia was defined as a value of serum calcium (Ca) greater than or equal to 10.3 mg/dL.
  Hyperphosphatemia was defined as a value of serum phosphorus (P) greater than or equal to 5.5 mg/dL.
  Elevated Ca×P was defined as as greater or equal to 56.65 mg^2/dL^2, calculated as the result of multiplying the maximum values of calcium (10.3 mg/dL) and phosphorus (5.5 mg/dL).
Time Frame: Baseline Week 1 (Study Visit 1), Week 12 (Study Visit 3), Week 24 (Final Study Visit)
Population: Participants with valid assessments at given time point.
Measure: Number; unit: percentage of participants
Groups:
- Paricalcitol IV: Baseline: Baseline Visit: Participants with a diagnosis of chronic kidney disease stage V undergoing hemodialysis were treated with paricalcitol IV per routine clinical practice, according to prescribing information approved in Venezuela and clinical criteria.
- Paricalcitol IV: Week 12: Week 12 Visit: Participants with a diagnosis of chronic kidney disease stage V undergoing hemodialysis were treated with paricalcitol IV per routine clinical practice, according to prescribing information approved in Venezuela and clinical criteria.
- Paricalcitol IV: Week 24: Week 24 Visit: Participants with a diagnosis of chronic kidney disease stage V undergoing hemodialysis were treated with paricalcitol IV per routine clinical practice, according to prescribing information approved in Venezuela and clinical criteria.
Arm/Group | Paricalcitol IV: Baseline | Paricalcitol IV: Week 12 | Paricalcitol IV: Week 24
Number analyzed (Participants) | 105 | 70 | 50
percentage of participants
  Hypercalcemia | 1.90 | 1.42 | 14.00
  Hyperphosphatemia | 28.57 | 42.85 | 38.00
  Elevations of (Ca x P) | 15.23 | 32.85 | 20.00

3. Secondary Outcome: Number of Participants Achieving Parathyroid Hormone (PTH) Levels < 300 pg/mL
Description: Participants who achieved PTH Levels < 300 pg/mL between the first and third study visit (Baseline to Week 12) and the third and final study visit (Week 12 to Week 24).
Time Frame: Baseline to Week 12, Week 12 to Week 24
Population: All participants; n=participants with valid PTH values at given time point.
Measure: Number; unit: participants
Arm/Group | Paricalcitol IV
Number analyzed (Participants) | 105
participants
  Baseline to Week 12; n=70 | 14
  Week 12 to Week 24; n=50 | 14

4. Secondary Outcome: Number of Participants Achieving PTH Level Reductions to < 300 pg/mL or 30% Below Baseline in 12 or 24 Weeks
Description: Number of participants achieving PTH level reductions to < 300 pg/mL or 30% below Baseline in 12 weeks (Baseline to Week 12 or Week 12 to Week 24) or in 24 weeks (Baseline to Week 24).
Time Frame: Baseline Week 1 (Study Visit 1) to Week 24 (Final Study Visit)
Population: All participants; n=number of participants with valid PTH values at given time point.
Measure: Number; unit: participants
Arm/Group | Paricalcitol IV
Number analyzed (Participants) | 105
participants
  Baseline to Week 12 (12 weeks); n=70 | 14
  Week 12 to Week 24 (12 weeks); n=50 | 13
  Baseline to Week 24 (24 weeks); n=50 | 16

5. Secondary Outcome: European Quality of Life 5 Dimensions (EQ-5D) Parameters of Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression At Baseline, Week 12, and Week 24
Description: The EQ-5D questionnaire is an international, standardized, generic instrument for describing and valuing health status that is divided into 5 parameters that include mobility, self-care, usual activities, pain/discomfort, anxiety/depression and a visual analogue scale (VAS). For each parameter other than the VAS, participants are asked to indicate which of 5 statements (from 'no problem' to 'extreme problem') best describes their health state.
Time Frame: Baseline Week 1 (Study Visit 1), Week 12 (Study Visit 3), Week 24 (Final Study Visit)
Population: Participants with valid assessments at given time point.
Measure: Number; unit: participants
Arm/Group | Paricalcitol IV: Baseline | Paricalcitol IV: Week 12 | Paricalcitol IV: Week 24
Number analyzed (Participants) | 104 | 70 | 50
participants
  Mobility: No Problems | 64 | 36 | 27
  Mobility: Slight Problems | 13 | 15 | 13
  Mobility: Moderate Problems | 13 | 6 | 8
  Mobility: Severe Problems | 5 | 3 | 2
  Mobility: Unable to Walk About | 1 | 0 | 0
  Mobility: Unknown | 8 | 10 | 0
  Self-Care: No Problems | 80 | 50 | 40
  Self-Care: Slight Problems | 8 | 3 | 7
  Self-Care: Moderate Problems | 5 | 3 | 3
  Self-Care: Severe Problems | 0 | 3 | 0
  Self-Care: Unable to Wash or Dress Self | 3 | 1 | 0
  Self-Care: Unknown | 8 | 10 | 0
  Usual Activities: No Problems | 53 | 37 | 28
  Usual Activities: Slight Problems | 26 | 13 | 15
  Usual Activities: Moderate Problems | 9 | 6 | 5
  Usual Activities: Severe Problems | 5 | 2 | 1
  Usual Activities: Unable to Do Usual Activities | 3 | 2 | 1
  Usual Activities: Unknown | 8 | 10 | 0
  Pain/Discomfort: None | 39 | 30 | 21
  Pain/Discomfort: Slight | 41 | 20 | 18
  Pain/Discomfort: Moderate | 13 | 9 | 10
  Pain/Discomfort: Severe | 2 | 1 | 1
  Pain/Discomfort: Extreme | 2 | 0 | 0
  Pain/Discomfort: Unknown | 7 | 10 | 0
  Anxiety/Depression: None | 66 | 46 | 39
  Anxiety/Depression: Slight | 24 | 11 | 9
  Anxiety/Depression: Moderate | 4 | 2 | 2
  Anxiety/Depression: Severe | 3 | 0 | 0
  Anxiety/Depression: Extreme | 0 | 0 | 0
  Anxiety/Depression: Unknown | 7 | 11 | 0

6. Secondary Outcome: European Quality of Life 5 Dimensions (EQ-5D) Visual Analogue Scale (VAS) Scores At Baseline, Week 12, and Week 24
Description: The EQ-5D questionnaire is an international, standardized, generic instrument for describing and valuing health status that is divided into 5 parameters that include mobility, self-care, usual activities, pain/discomfort, anxiety/depression and a VAS. For the VAS portion, health status is assessed by participants on a vertical, visual analog scale from 0 to 100 where the endpoints are labeled 'worst imaginable health state' (0) and 'best imaginable health state' (100).
Time Frame: Baseline Week 1 (Study Visit 1), Week 12 (Study Visit 3), Week 24 (Final Study Visit)
Population: Participants with valid assessments at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paricalcitol IV: Baseline | Paricalcitol IV: Week 12 | Paricalcitol IV: Week 24
Number analyzed (Participants) | 94 | 59 | 48
units on a scale | 77.98 (16.21) | 84.31 (14.52) | 80.33 (18.28)

7. Secondary Outcome: Beck Depression Inventory (BDI) Scores At Baseline and Final Study Visit
Description: BDI is a 21-item questionnaire, participant self-report rating inventory that measures characteristic attitudes and symptoms of depression. The range of scores is 0 to 63, with a higher value representing a worse outcome.
Time Frame: Baseline Week 1 (Study Visit 1), Week 24 (Final Study Visit)
Population: Participants with a complete, valid assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paricalcitol IV: Baseline | Paricalcitol IV: Week 24
Number analyzed (Participants) | 88 | 45
units on a scale | 10.39 (7.04) | 7.96 (5.75)

ADVERSE EVENTS:
Time Frame: From time of informed consent until 30 days or 5 half-lives following intake of the last dose of physician-prescribed treatment.
Arm/Group | Paricalcitol IV
Serious Adverse Events (participants affected / at risk) | 9/105
Other Adverse Events (participants affected / at risk) | 21/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol IV (N=105)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Parathyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Sepsis (Infections and infestations) | 2
Spinal cord compression (Musculoskeletal and connective tissue disorders) | 1
Drowning (Social circumstances) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol IV (N=105)
Gastritis (Gastrointestinal disorders) | 6
Insomnia (Nervous system disorders) | 4
Neuropathic pain (Nervous system disorders) | 2
Catheter related infection (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Pain in extremities (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain (General disorders) | 1
Chest pain (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.